CLINICAL TRIAL: NCT04109690
Title: A Phase I-II Study of a Liposomal Formulation of Cytarabine and Daunorubicin (CPX-351) in Patients Treated for Higher-risk Myelodysplastic Syndromes Experiencing Hypomethylating Agent Failure.
Brief Title: CPX-351 in Patients Treated for Higher-risk Myelodysplastic Syndromes Experiencing Hypomethylating Agent Failure.
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Failure to enroll
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000024262
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: MDS
Keywords: MDS
MeSH Terms: interventions — CPX-351

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPX-351 (Experimental): Phase I will evaluate the safety and tolerability of CPX-351 (44mg/m2 of daunorubicin and 100mg/m2 of cytarabine) administered on 2 days (day 1 and day 5) to determine the Phase II dose. Phase II will evaluate the efficacy of the RP2D.
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — Patients in both Phase I and II can receive a maximum of two induction and six consolidation cycles on an inpatient or outpatient basis per local hospital standard of care.

SUMMARY:
The proposed study is of a Liposomal formulation of cytarabine and daunorubicin (CPX-351) in patients treated for higher-risk myelodysplastic syndromes (MDS) experiencing hypomethylating agent failure.

DETAILED DESCRIPTION:
Proposed is a two-phase study. The Phase I portion will confirm the tolerability and safety of CPX-351 chemotherapy. Patients who meet eligibility criteria will receive dose level 1 of CPX-351 (44mg/m2 of daunorubicin and 100mg/m2 of cytarabine) on 2 days (day 1 and day 5) of the cycle.

If less than 2 dose limiting toxicity (DLT) are observed in the first cohort of 6, we will increase level of exposure to Dose Level 2 by giving (44mg/m2 of daunorubicin and 100mg/m2 of cytarabine) on days 1, 3 and 5 of

* If less than 2 DLTs are observed Dose Level 2 will become the Recommended Phase II dose (RP2D)
* If 2 or more DLTs are observed Dose Level 1 will become the RP2D If 2 or more DLTs are observed in the first cohort of 6 patients, another 6 patients will be enrolled at dose level -1 (29mg/m2 of daunorubicin and 65mg/m2 of cytarabine) on day 1 and 5.
* If less than 2 DLTs are observed Dose Level -1 will become the RP2D
* If 2 or more patients experience a DLT at dose -1 the study will be stopped Patients failing to achieve a response after cycle 1 will be offered a second cycle of induction with for dose level 1 and 2 (44mg/m2 of daunorubicin and 100mg/m2 of cytarabine) on day 1 and 5 of induction 2. And for dose level-1, (29mg/m2 of daunorubicin and 65mg/m2 of cytarabine) on day 1 and 5 of induction 2.

Phase II: Once the RP2D is confirmed we will enroll 12 patients. If 3 or more responses are observed an additional 12 patients will be enrolled for a total of 24. If 7 out of 24 evaluable patients achieve response, an additional 24 patients will be enrolled for a total of 48 patients.

• If less than 3 responses are observed in the first 12 patients, the study will be terminated.

The outcomes presented in this protocol are associated with the Phase II of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of MDS o (according to World Health Organization 2016 classification) made prior to administration off HMA
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2
* Patient must have recovered from toxicities of any prior treatment regimen (no CTCAE grading over 1 for non-hematological toxicities and a return to baseline for hematological values)
* Patient is considered eligible for chemotherapy (at discretion of local investigator)
* Patient must have been treated with a hypomethylating agent (+/- other agents) and

  * be treated for at least 4 cycles (16 weeks) and have a stable marrow disease (no response) or
  * progressed without prior response based on MDS International Working Group (IWG) 2006 response criteria or
  * relapsed after an initial response based on MDS IWG 2006 response criteria.
* Adequate liver and renal function:

  * Estimated creatinine clearance above 40 ml/min
  * Total bilirubin ≤ 1.5 x the Upper Limit of Normal (ULN) or ≤ 3.0 x the ULN unless considered due to Gilbert's syndrome,
  * Alanine aminotransferase (ALT) (SGPT), and aspartate aminotransferase (AST) (SGOT) ≤ 2.5 x the ULN. For patients with hepatic leukemic involvement Alanine aminotransferase (ALT) (SGPT), and aspartate aminotransferase (AST) (SGOT) ≤ 5.0 x the ULN t
* Able to understand and sign the written informed consent
* Serum or urine pregnancy test (for female patients of childbearing potential) with a minimum sensitivity of 25 IU/L or equivalent units of human chorionic gonadotropin (HCG) negative at screening.
* Males and female patients both of childbearing potential and at risk for pregnancy must agree to use two highly effective method(s) of contraception throughout the study and for 180 days after the last dose of CPX-351 whichever occurs later.
* Female patients who are not of childbearing potential (i.e. meet at least 1 of the following criteria):

  * Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  * Have medically confirmed ovarian failure;
  * Have achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by having a serum follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal women.

Exclusion Criteria:

* Any prior induction chemotherapy (defined as treatment with standard or high dose cytarabine in combination with an anthracycline and/or other agents)
* Any investigational agent administered within a month prior to inclusion or within 5 half-lives of the investigational agent whichever is longer.
* Promyelocytic acute leukemia and core binding factor acute leukemia.
* Active Central nervous system (CNS) disease
* Any severe chronic disease potentially interfering with the protocol including HIV infection, active or chronic hepatitis B or C. Testing will be completed during screening period.
* Any significant social condition that could limit the understanding of the study or the compliance to the protocol including but not limited to severe or uncontrolled psychiatric illness.
* Any sign of active uncontrolled disease including but not restricted to cardiac disease, infections and platelet refractoriness.
* Any other malignancy with active treatment within the past 1 year other than basal cell skin cancer or carcinoma in situ of the cervix.
* New York Heart Association (NYHA) grade 3 or 4 cardiac failure, or left ventricular ejection fraction (LVEF) below 50%
* Patients who have received a cumulative dose of anthracyclines superior to a total of 300mg/m2 of daunorubicin in the absence of prior mediastinal radiation or 150mg/m2 if the patient had a prior mediastinal radiation
* Oxygen dependency as defined by a chronic need of oxygen at least 2l/min for at least 6h a day.
* Women who are pregnant, planning to become pregnant, or who are currently breastfeeding
* Persistence of any clinically relevant (CTCAE grade 2 or above) toxicities from previous therapy
* Any other condition that, according to the investigator, may forbid the administration of CPX-351
* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or another copper-metabolism disorder
* Major injuries and/or surgery within the past 4 weeks prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 24 months
  The Phase II primary objective is to determine the overall response rate (CR/CRi) of CPX-351 in MDS patients experiencing hypomethylation (HMA) failure.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Prebet, MD, PHD, Principal Investigator — Yale University
Locations (1):
- Yale University; Smilow Cancer Center, New Haven, Connecticut, United States